CLINICAL TRIAL: NCT06543589
Title: A Randomised Trial Comparing of High Flow Nasal Cannula Versus Cpap for Initial Respiratory Stabilisation of Very Premature Infants
Brief Title: Comparing of High Flow Nasal Cannula Versus Cpap for Initial Respiratory Stabilisation of Very Premature Infants
Acronym: SIMPLSAFE3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jonáš Klára, Investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 8/24
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-08

CONDITIONS: Premature; Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: The randomization unit in this study is the center, rather than individual patients. Centers will be randomized to either the ARM A or ARM B at each time period using a stepped-wedge cluster-randomized design. A randomization schedule will be generated using a computer-based random number generator to ensure unbiased allocation. At each of the specified time periods, a random subset of centers will be selected to switch from control to intervention.
  While it is not feasible to blind the centers to their intervention status due to the nature of the study, the data analysts will be blinded to the group assignments to minimize bias. The randomization will be implemented by the study coordinator, who will notify each center of their assignment at the beginning of each time period. This approach ensures that each center will eventually receive the intervention, allowing for both within-center and between-center comparisons, thus enhancing the robustness of the study findings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A (CPAP group) (No Intervention): Infants randomized to the ARM A group will be stabilized on CPAP, according to the standard procedure of each participating center.
- ARM B (HFNC group) (Experimental): For infants randomly assigned to the ARM B group, the respiratory support will be provided by devices that deliver a blend of heated and humidified gas mixture of air and oxygen at gas flows exceeding 8 L/ min via binasal cannula.
  Interventions: Device: High-flow-nasal-cannula

INTERVENTIONS:
Device: High-flow-nasal-cannula — Respiratory support will be provided by devices that deliver a blend of heated and humidified gas mixture of air and oxygen at gas flows exceeding 8 L/ min via binasal cannula.
  Arms: ARM B (HFNC group)

SUMMARY:
Non-invasive continuous positive airway pressure (CPAP) stabilizes premature newborns, but its optimal pressure is unknown. High-flow nasal cannula (HFNC) is an alternative that minimizes trigeminal stimulation but lacks precise pressure control. Initial studies show HFNC's feasibility and effectiveness. This study hypothesizes that HFNC can deliver adequate pressure, reduce the need for positive pressure ventilation, and support safe stabilization of very premature infants. The trial compares the effectiveness and safety of HFNC versus CPAP in the delivery room and during transport to the neonatal intensive care unit in very premature infants. The primary objective is to compare HFNC and CPAP in reducing the need for positive pressure ventilation in very premature infants immediately after birth. The study includes very premature infants delivered between 28+0 and 31+6 weeks gestation in 10 tertiary referral centers (nine in the Czech Republic, one in Slovakia). Approximately 443 patients are required to detect a 15% relative decrease in the need for positive pressure ventilation between trial groups. Centers will be randomized to either CPAP or HFNC at each time period, with parental consent obtained before birth. The primary endpoint is the proportion of neonates requiring positive pressure ventilation within the first 10 minutes post-birth.

DETAILED DESCRIPTION:
Background and Rationale

The stabilization of very premature infants (VPIs) immediately after birth is crucial, as their underdeveloped lungs are prone to respiratory distress. Non-invasive continuous positive airway pressure (CPAP) is commonly recommended in the delivery room and during transport to the NICU. While CPAP can help maintain airway pressure and support spontaneous breathing, its optimal pressure settings are not yet established. Furthermore, when CPAP pressure is increased for infants who are not breathing spontaneously, it often necessitates positive pressure ventilation (PPV), which may lead to lung injury and increase the risk of complications.

CPAP's reliance on a face mask requires frequent adjustments, which can trigger reflexes that may exacerbate bradycardia, potentially destabilizing the neonate. High-flow nasal cannula (HFNC) offers an alternative that reduces direct facial stimulation, thus potentially lowering the occurrence of these reflex-induced events. Preliminary studies suggest that HFNC is both feasible and effective in supporting some premature infants, though HFNC does not provide the precise pressure control seen with CPAP. This study is designed to evaluate if HFNC can provide effective airway pressure for initial lung clearance, decrease the need for PPV, and support safe respiratory stabilization of VPIs immediately after birth.

Hypothesis

HFNC will reduce upper airway resistance and deliver adequate positive pressure for lung aeration in spontaneously breathing, very immature neonates. Compared to CPAP, HFNC's reduced physical stimulation may decrease the requirement for PPV, promoting a smoother transition to stable lung function and cardiopulmonary stabilization in very preterm infants.

Trial Aim

This trial aims to compare the effectiveness and safety of HFNC and CPAP in stabilizing severely premature neonates in the delivery room and during transport to the NICU. The primary endpoint is the proportion of neonates requiring PPV within the first 10 minutes post-birth, to determine if HFNC can reduce the need for PPV more effectively than CPAP.

Objectives

The primary objective is to evaluate whether HFNC can reduce the need for PPV compared to CPAP in very premature infants immediately after birth. Secondary objectives will focus on achieving specific oxygenation and ventilation milestones without PPV, including SpO₂ levels and FiO₂ requirements.

Study Design

This is a stepped-wedge cluster randomized controlled trial (RCT) involving 10 tertiary perinatal care centers (9 in the Czech Republic, 1 in Slovakia). Participating centers will switch between using HFNC and CPAP during specified time periods. Randomization will determine the order in which each center uses either HFNC or CPAP across six to ten periods of approximately 90 days each.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth between 28+0 and 31+6 weeks by the best obstetric estimate.
* Written informed consent from parent/legal guardian(s) is obtained before delivery.

Exclusion Criteria:

* Peripartal hypoxia with pH < 7,1
* Significant congenital malformations.
* IUGR with estimated weight of fetus below 800g.
* Condition that has an adverse effect on breathing/ventilation or oxygenation, including congenital diaphragmatic hernia, trachea-oesophageal fistula, cyanotic heart disease and surfactant protein deficiency.
* Documented decision to give palliative neonatal care.

Ages: 1 Minute to 5 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 443 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Positive pressure ventilation (PPV) | 10 minutes after delivery
  The primary endpoint of the trial is to demonstrate a difference in the proportion of neonates requiring PPV administration in the delivery room during the first 10 minutes post-birth.
  This will be recorded as a binary outcome (yes/no) indicating whether PPV was administered. Each neonate's need for PPV should be documented by the clinical team and recorded in a standardized data collection form immediately after delivery.

SECONDARY OUTCOMES:
SpO2 >80% within the first 5 minutes of life | 5 minutes after delivery
  Achieving SpO2 >80% within the first 5 minutes of life, regardless of FiO2 without the need of PPV administration.
  Oxygen saturation (SpO₂) will be measured continuously using a pulse oximeter attached to the infant.
SpO2 >90% with FiO2 ≤ 0.40 within the first 10 minutes of life | 10 minutes after delivery
  Achieving SpO2 >90% with FiO2 ≤ 0.40 within the first 10 minutes of life without the need for PPV.
  Oxygen saturation (SpO₂) will be measured continuously using a pulse oximeter attached to the infant.
Stabilization on selected ventilatory support | 3 hours after delivery
  Stabilization on selected ventilatory support with FiO2 ≤ 0.35 without the use of PPV at 3h of life.
  FiO₂ and respiratory support (CPAP or HFNC) will be documented.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madar J, Roehr CC, Ainsworth S, Ersdal H, Morley C, Rudiger M, Skare C, Szczapa T, Te Pas A, Trevisanuto D, Urlesberger B, Wilkinson D, Wyllie JP. European Resuscitation Council Guidelines 2021: Newborn resuscitation and support of transition of infants at birth. Resuscitation. 2021 Apr;161:291-326. doi: 10.1016/j.resuscitation.2021.02.014. Epub 2021 Mar 24. PMID 33773829
- [Background] Kirpalani H, Ratcliffe SJ, Keszler M, Davis PG, Foglia EE, Te Pas A, Fernando M, Chaudhary A, Localio R, van Kaam AH, Onland W, Owen LS, Schmolzer GM, Katheria A, Hummler H, Lista G, Abbasi S, Klotz D, Simma B, Nadkarni V, Poulain FR, Donn SM, Kim HS, Park WS, Cadet C, Kong JY, Smith A, Guillen U, Liley HG, Hopper AO, Tamura M; SAIL Site Investigators. Effect of Sustained Inflations vs Intermittent Positive Pressure Ventilation on Bronchopulmonary Dysplasia or Death Among Extremely Preterm Infants: The SAIL Randomized Clinical Trial. JAMA. 2019 Mar 26;321(12):1165-1175. doi: 10.1001/jama.2019.1660. PMID 30912836
- [Background] Lista G, Cavigioli F, La Verde PA, Castoldi F, Bresesti I, Morley CJ. Effects of Breathing and Apnoea during Sustained Inflations in Resuscitation of Preterm Infants. Neonatology. 2017;111(4):360-366. doi: 10.1159/000454799. Epub 2017 Jan 25. PMID 28118641
- [Background] Martherus T, Oberthuer A, Dekker J, Hooper SB, McGillick EV, Kribs A, Te Pas AB. Supporting breathing of preterm infants at birth: a narrative review. Arch Dis Child Fetal Neonatal Ed. 2019 Jan;104(1):F102-F107. doi: 10.1136/archdischild-2018-314898. Epub 2018 Jul 26. PMID 30049727
- [Background] Kuypers K, Martherus T, Lamberska T, Dekker J, Hooper SB, Te Pas AB. Reflexes that impact spontaneous breathing of preterm infants at birth: a narrative review. Arch Dis Child Fetal Neonatal Ed. 2020 Nov;105(6):675-679. doi: 10.1136/archdischild-2020-318915. Epub 2020 Apr 29. PMID 32350064
- [Background] Kuypers KLAM, Hopman A, Cramer SJE, Dekker J, Visser R, Hooper SB, Te Pas AB. Effect of initial and subsequent mask applications on breathing and heart rate in preterm infants at birth. Arch Dis Child Fetal Neonatal Ed. 2023 Nov;108(6):594-598. doi: 10.1136/archdischild-2022-324835. Epub 2023 Apr 20. PMID 37080734
- [Background] Reynolds P, Leontiadi S, Lawson T, Otunla T, Ejiwumi O, Holland N. Stabilisation of premature infants in the delivery room with nasal high flow. Arch Dis Child Fetal Neonatal Ed. 2016 Jul;101(4):F284-7. doi: 10.1136/archdischild-2015-309442. Epub 2016 Jan 5. PMID 26733541
- [Background] Siva NV, Reynolds PR. Stabilisation of the preterm infant in the delivery room using nasal high flow: A 5-year retrospective analysis. Acta Paediatr. 2021 Jul;110(7):2065-2071. doi: 10.1111/apa.15824. Epub 2021 Mar 8. PMID 33638878
- [Background] Roberts CT, Hodgson KA. Nasal high flow treatment in preterm infants. Matern Health Neonatol Perinatol. 2017 Sep 6;3:15. doi: 10.1186/s40748-017-0056-y. eCollection 2017. PMID 28904810
- [Background] Mazmanyan P, Darakchyan M, Pinkham MI, Tatkov S. Mechanisms of nasal high flow therapy in newborns. J Appl Physiol (1985). 2020 Apr 1;128(4):822-829. doi: 10.1152/japplphysiol.00871.2019. Epub 2020 Feb 20. PMID 32078463
- [Background] Bjorland PA, Oymar K, Ersdal HL, Rettedal SI. Incidence of newborn resuscitative interventions at birth and short-term outcomes: a regional population-based study. BMJ Paediatr Open. 2019 Dec 29;3(1):e000592. doi: 10.1136/bmjpo-2019-000592. eCollection 2019. PMID 31909225
- [Background] Roberts CT, Owen LS, Manley BJ, Froisland DH, Donath SM, Dalziel KM, Pritchard MA, Cartwright DW, Collins CL, Malhotra A, Davis PG; HIPSTER Trial Investigators. Nasal High-Flow Therapy for Primary Respiratory Support in Preterm Infants. N Engl J Med. 2016 Sep 22;375(12):1142-51. doi: 10.1056/NEJMoa1603694. PMID 27653564
- [Background] Manley BJ, Arnolda GRB, Wright IMR, Owen LS, Foster JP, Huang L, Roberts CT, Clark TL, Fan WQ, Fang AYW, Marshall IR, Pszczola RJ, Davis PG, Buckmaster AG; HUNTER Trial Investigators. Nasal High-Flow Therapy for Newborn Infants in Special Care Nurseries. N Engl J Med. 2019 May 23;380(21):2031-2040. doi: 10.1056/NEJMoa1812077. PMID 31116919